CLINICAL TRIAL: NCT02081807
Title: Sequential Expansion of Comparative Effectiveness of Oral Anticoagulants: A Cohort Study
Brief Title: Sequential Expansion of Comparative Effectiveness of Anticoagulants
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160.207
Record Dates: First submitted 2014-03-06; First posted 2014-03-07 (Estimated); Results first posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Dabigatran
- Warfarin

SUMMARY:
This cohort study is the sequential expansion of the comparative effectiveness study of oral anticoagulants and plans to identify initiators of oral anticoagulants using electronic claims data from a commercial insurance database to quantify associations between anticoagulant choice (warfarin and dabigatran) and the occurrence of selected outcomes in patients with non-valvular atrial fibrillation at risk for stroke.

ELIGIBILITY:
Inclusion criteria:

* A recorded diagnosis of atrial fibrillation.
* Initiation of anticoagulant medication (dabigatran (or other new oral anticoagulants as they become available) or warfarin).
* At least 18 years of age on the date of anticoagulant initiation.
* Congestive Heart Failure, Hypertension, Age > 75, Diabetes Mellitus, Prior Stroke or Transient Ischemic Attack, Vascular Disease, Age 65-74, Sex Category (CHA2DS2-VASc) score at least 1

Exclusion criteria:

* Patients with missing or ambiguous age or sex information.
* Patients with evidence of valvular disease.
* Patients with less than 12 months enrolment preceding the date of anticoagulant initiation
* Patients with a dispensing of any oral anticoagulant during the 12 months preceding the date of anticoagulant initiation
* Patients with a nursing home stay during the 12 months preceding the date of anticoagulant initiation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years of age and older with non-valvular AF initiating oral anticoagulation therapy
Sampling Method: Non-Probability Sample
Enrollment: 221228 (Actual)
Dates: Start 2014-03-07 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data for the patients included in this cohort study arose from two de-identified research databases, US MarketScan and Optum Research Database
Pre-assignment Details: In this non-interventional study based on existing data, no patients were screened.
Groups:
- Optum Clinformatics - Dabigatran: Patients with non- valvular atrial fibrillation (NVAF) and new initiators of dabigatran, during October 2010 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database before treatment initiation
- Optum Clinformatics - Warfarin: Patients with non- valvular atrial fibrillation (NVAF) and new initiators of warfarin, during October 2010 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database before treatment initiation
- Optum Clinformatics - Rivaroxaban: Patients with non- valvular atrial fibrillation (NVAF) and new initiators of rivaroxaban, during July 2011 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database before treatment initiation
- Optum Clinformatics - Apixaban: Patients with non- valvular atrial fibrillation (NVAF) and new initiators of apixaban, during January 2013 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database before treatment initiation
- MarketScan - Dabigatran: Patients with non- valvular atrial fibrillation (NVAF) and new initiators of dabigatran, during October 2010 to September 2015 who were enrolled for a minimum of 12 months in MarketScan before treatment initiation
- MarketScan - Warfarin: Patients with non- valvular atrial fibrillation (NVAF) and new initiators of warfarin, during October 2010 to September 2015 who were enrolled for a minimum of 12 months in MarketScan before treatment initiation
- MarketScan - Rivaroxaban: Patients with non- valvular atrial fibrillation (NVAF) and new initiators of rivaroxaban, during July 2011 to September 2015 who were enrolled for a minimum of 12 months in MarketScan before treatment initiation
- MarketScan - Apixaban: Patients with non- valvular atrial fibrillation (NVAF) and new initiators of apixaban, during January 2013 to September 2015 who were enrolled for a minimum of 12 months in MarketScan before treatment initiation
Period: Overall Study
Arm/Group | Optum Clinformatics - Dabigatran | Optum Clinformatics - Warfarin | Optum Clinformatics - Rivaroxaban | Optum Clinformatics - Apixaban | MarketScan - Dabigatran | MarketScan - Warfarin | MarketScan - Rivaroxaban | MarketScan - Apixaban
Started | 7668 | 26149 | 14852 | 9112 | 27456 | 76055 | 40207 | 19729
Completed | 7668 | 26149 | 14852 | 9112 | 27456 | 76055 | 40207 | 19729
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Patients with non- valvular atrial fibrillation (NVAF) and new initiators of dabigatran, warfarin, rivaroxaban or apixaban during October 2010 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database or MarketScan before treatment initiation
Groups:
- Total: Total of all reporting groups
Arm/Group | Optum Clinformatics - Dabigatran | Optum Clinformatics - Warfarin | Optum Clinformatics - Rivaroxaban | Optum Clinformatics - Apixaban | MarketScan - Dabigatran | MarketScan - Warfarin | MarketScan - Rivaroxaban | MarketScan - Apixaban | Total
Number analyzed (Participants) | 7668 | 26149 | 14852 | 9112 | 27456 | 76055 | 40207 | 19729 | 221228
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (11.3) | 69.9 (11.8) | 68.0 (11.9) | 71.9 (11.2) | 67.1 (12.1) | 71.0 (12.1) | 67.6 (12.2) | 69.4 (12.3) | 69.2 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2315 | 10143 | 5483 | 3911 | 9774 | 29693 | 15014 | 7747 | 84080
  Male | 5353 | 16006 | 9369 | 5201 | 17682 | 46362 | 25193 | 11982 | 137148
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Stroke (Hemorrhagic, Ischemic, or Stroke of Uncertain Classification)
Description: The rate of overall stroke (hemorrhagic, ischemic or stroke of uncertain classification ) in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. The outcome definition includes following: As primary International Classification of Diseases, Ninth Revision (ICD-9) discharge diagnosis (Dx): 431.x Intracerebral hemorrhage (ICH), 433.x1 Occlusion and stenosis of precerebral arteries with cerebral infarction, 434.x1 Occlusion and stenosis of cerebral arteries with cerebral infarction, 436.x Acute, but ill-defined cerebrovascular events.
Time Frame: From October 2010 to September 2015 (the study period)
Population: Patients with non-valvular atrial fibrillation (NVAF) and new initiators of dabigatran and warfarin during October 2010 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database or MarketScan before treatment initiation and matched on propensity scores (PS). Primary analysis represented an 'as treated' approach.
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Groups:
- Optum Clinformatics - Dabigatran vs. Warfarin (Dabigatran): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of dabigatran, during October 2010 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database before treatment initiation and matched on propensity scores with warfarin
- Optum Clinformatics - Dabigatran vs. Warfarin (Warfarin): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of warfarin, during October 2010 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database before treatment initiation and matched on propensity scores with dabigatran
- MarketScan - Dabigatran vs. Warfarin (Dabigatran): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of dabigatran, during October 2010 to September 2015 who were enrolled for a minimum of 12 months in MarketScan before treatment initiation and matched on propensity scores with warfarin
- MarketScan - Dabigatran vs. Warfarin (Warfarin): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of warfarin, during October 2010 to September 2015 who were enrolled for a minimum of 12 months in MarketScan before treatment initiation and matched on propensity scores with dabigatran
- Optum Clinformatics - Rivaroxaban vs. Warfarin (Rivaroxaban): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of rivaroxaban, during July 2011 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database before treatment initiation and matched on propensity scores with warfarin
- Optum Clinformatics - Rivaroxaban vs. Warfarin (Warfarin): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of warfarin, during July 2011 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database before treatment initiation and matched on propensity scores with rivaroxaban
- MarketScan - Rivaroxaban vs. Warfarin (Rivaroxaban): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of rivaroxaban, during July 2011 to September 2015 who were enrolled for a minimum of 12 months in MarketScan before treatment initiation and matched on propensity scores with warfarin
- MarketScan - Rivaroxaban vs. Warfarin (Warfarin): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of warfarin, during July 2011 to September 2015 who were enrolled for a minimum of 12 months in MarketScan before treatment initiation and matched on propensity scores with rivaroxaban
- Optum Clinformatics - Apixaban vs. Warfarin (Apixaban): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of apixaban, during January 2013 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database before treatment initiation and matched on propensity scores with warfarin
- Optum Clinformatics - Apixaban vs. Warfarin (Warfarin): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of warfarin, during January 2013 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database before treatment initiation and matched on propensity scores with apixaban
- MarketScan - Apixaban vs. Warfarin (Apixaban): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of apixaban, during January 2013 to September 2015 who were enrolled for a minimum of 12 months in MarketScan before treatment initiation and matched on propensity scores with warfarin
- MarketScan - Apixaban vs. Warfarin (Warfarin): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of warfarin, during January 2013 to September 2015 who were enrolled for a minimum of 12 months in MarketScan before treatment initiation and matched on propensity scores with apixaban
Arm/Group | Optum Clinformatics - Dabigatran vs. Warfarin (Dabigatran) | Optum Clinformatics - Dabigatran vs. Warfarin (Warfarin) | MarketScan - Dabigatran vs. Warfarin (Dabigatran) | MarketScan - Dabigatran vs. Warfarin (Warfarin) | Optum Clinformatics - Rivaroxaban vs. Warfarin (Rivaroxaban) | Optum Clinformatics - Rivaroxaban vs. Warfarin (Warfarin) | MarketScan - Rivaroxaban vs. Warfarin (Rivaroxaban) | MarketScan - Rivaroxaban vs. Warfarin (Warfarin) | Optum Clinformatics - Apixaban vs. Warfarin (Apixaban) | Optum Clinformatics - Apixaban vs. Warfarin (Warfarin) | MarketScan - Apixaban vs. Warfarin (Apixaban) | MarketScan - Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 6125 | 6125 | 23323 | 23323 | 10373 | 10373 | 25147 | 25147 | 7065 | 7065 | 12523 | 12523
Incidence rate per 100 person-years | 0.90 [0.60 to 1.30] | 1.01 [0.66 to 1.50] | 0.64 [0.51 to 0.80] | 0.99 [0.80 to 1.20] | 0.80 [0.56 to 1.11] | 1.02 [0.72 to 1.39] | 0.78 [0.64 to 0.94] | 1.09 [0.90 to 1.31] | 1.08 [0.74 to 1.53] | 1.26 [0.86 to 1.80] | 0.62 [0.44 to 0.84] | 1.16 [0.87 to 1.51]
Statistical Analysis 1: Comparison: Optum Clinformatics - Dabigatran vs. Warfarin (Dabigatran) vs Optum Clinformatics - Dabigatran vs. Warfarin (Warfarin); Optum Clinformatic-Dabigatran vs. Warfarin (as reference group); Test type: Other; Regression, Cox; Cox proportional-hazards regression analysis was used to compute Hazard ratios (HR) and corresponding 95% confidence intervals (CI); Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.57 to 1.76]
Statistical Analysis 2: Comparison: MarketScan - Dabigatran vs. Warfarin (Dabigatran) vs MarketScan - Dabigatran vs. Warfarin (Warfarin); MarketScan-Dabigatran vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.52 to 0.94]
Statistical Analysis 3: Comparison: Optum Clinformatics - Dabigatran vs. Warfarin (Dabigatran) vs Optum Clinformatics - Dabigatran vs. Warfarin (Warfarin) vs MarketScan - Dabigatran vs. Warfarin (Dabigatran) vs MarketScan - Dabigatran vs. Warfarin (Warfarin); This is a pooled analysis involving data from both MarketScan and Optum databases. MarketScan and Optum Clinformatic-Dabigatran vs. Warfarin (as reference group); Test type: Other; Regression, Cox; Cox proportional-hazards regression analysis was used to compute pooled HR and corresponding 95% CI using fixed effect meta-analysis; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.58 to 0.98]
Statistical Analysis 4: Comparison: Optum Clinformatics - Rivaroxaban vs. Warfarin (Rivaroxaban) vs Optum Clinformatics - Rivaroxaban vs. Warfarin (Warfarin); Optum Clinformatic- Rivaroxaban vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.53 to 1.35]
Statistical Analysis 5: Comparison: MarketScan - Rivaroxaban vs. Warfarin (Rivaroxaban) vs MarketScan - Rivaroxaban vs. Warfarin (Warfarin); MarketScan-Rivaroxaban vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.57 to 0.98]
Statistical Analysis 6: Comparison: Optum Clinformatics - Rivaroxaban vs. Warfarin (Rivaroxaban) vs Optum Clinformatics - Rivaroxaban vs. Warfarin (Warfarin) vs MarketScan - Rivaroxaban vs. Warfarin (Rivaroxaban) vs MarketScan - Rivaroxaban vs. Warfarin (Warfarin); This is a pooled analysis involving data from both MarketScan and Optum databases. MarketScan and Optum Clinformatic- Rivaroxaban vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.61 to 0.98]
Statistical Analysis 7: Comparison: Optum Clinformatics - Apixaban vs. Warfarin (Apixaban) vs Optum Clinformatics - Apixaban vs. Warfarin (Warfarin); Optum Clinformatic- Apixaban vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.53 to 1.51]
Statistical Analysis 8: Comparison: MarketScan - Apixaban vs. Warfarin (Apixaban) vs MarketScan - Apixaban vs. Warfarin (Warfarin); MarketScan-Apixaban vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.38 to 0.89]
Statistical Analysis 9: Comparison: Optum Clinformatics - Apixaban vs. Warfarin (Apixaban) vs Optum Clinformatics - Apixaban vs. Warfarin (Warfarin) vs MarketScan - Apixaban vs. Warfarin (Apixaban) vs MarketScan - Apixaban vs. Warfarin (Warfarin); This is a pooled analysis involving data from both MarketScan and Optum databases. MarketScan and Optum Clinformatic- Apixaban vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.50 to 0.96]

2. Primary Outcome: Major Bleeding
Description: The rate of major bleeding (Major intracranial bleeding and major extracranial bleed ) in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. For outcome definitions please refer the descriptions section of outcome 8 (major intracranial bleeding) and outcome 9 (major extracranial bleeding).
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Optum Clinformatics - Dabigatran vs. Warfarin (Dabigatran) | Optum Clinformatics - Dabigatran vs. Warfarin (Warfarin) | MarketScan - Dabigatran vs. Warfarin (Dabigatran) | MarketScan - Dabigatran vs. Warfarin (Warfarin) | Optum Clinformatics - Rivaroxaban vs. Warfarin (Rivaroxaban) | Optum Clinformatics - Rivaroxaban vs. Warfarin (Warfarin) | MarketScan - Rivaroxaban vs. Warfarin (Rivaroxaban) | MarketScan - Rivaroxaban vs. Warfarin (Warfarin) | Optum Clinformatics - Apixaban vs. Warfarin (Apixaban) | Optum Clinformatics - Apixaban vs. Warfarin (Warfarin) | MarketScan - Apixaban vs. Warfarin (Apixaban) | MarketScan - Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 6125 | 6125 | 23323 | 23323 | 10373 | 10373 | 25147 | 25147 | 7065 | 7065 | 12523 | 12523
Incidence rate per 100 person-years | 2.43 [1.91 to 3.05] | 5.23 [4.35 to 6.24] | 4.36 [4.00 to 4.74] | 6.06 [5.58 to 6.56] | 6.2 [5.5 to 7.0] | 6.3 [5.5 to 7.2] | 6.9 [6.5 to 7.4] | 7.5 [7.0 to 8.0] | 3.33 [2.69 to 4.07] | 6.83 [5.80 to 7.99] | 4.25 [3.74 to 4.80] | 7.96 [7.15 to 8.83]
Statistical Analysis 1: Comparison: Optum Clinformatics - Dabigatran vs. Warfarin (Dabigatran) vs Optum Clinformatics - Dabigatran vs. Warfarin (Warfarin); Optum Clinformatic-Dabigatran vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.38 to 0.69]
Statistical Analysis 2: Comparison: MarketScan - Dabigatran vs. Warfarin (Dabigatran) vs MarketScan - Dabigatran vs. Warfarin (Warfarin); MarketScan-Dabigatran vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.68 to 0.86]
Statistical Analysis 3: Comparison: Optum Clinformatics - Dabigatran vs. Warfarin (Dabigatran) vs Optum Clinformatics - Dabigatran vs. Warfarin (Warfarin) vs MarketScan - Dabigatran vs. Warfarin (Dabigatran) vs MarketScan - Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.72, 95% CI 2-sided [0.65 to 0.80]
Statistical Analysis 4: Comparison: Optum Clinformatics - Rivaroxaban vs. Warfarin (Rivaroxaban) vs Optum Clinformatics - Rivaroxaban vs. Warfarin (Warfarin); Optum Clinformatic- Rivaroxaban vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.88 to 1.26]
Statistical Analysis 5: Comparison: MarketScan - Rivaroxaban vs. Warfarin (Rivaroxaban) vs MarketScan - Rivaroxaban vs. Warfarin (Warfarin); MarketScan-Rivaroxaban vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.92 to 1.12]
Statistical Analysis 6: Comparison: Optum Clinformatics - Rivaroxaban vs. Warfarin (Rivaroxaban) vs Optum Clinformatics - Rivaroxaban vs. Warfarin (Warfarin) vs MarketScan - Rivaroxaban vs. Warfarin (Rivaroxaban) vs MarketScan - Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.94 to 1.12]
Statistical Analysis 7: Comparison: Optum Clinformatics - Apixaban vs. Warfarin (Apixaban) vs Optum Clinformatics - Apixaban vs. Warfarin (Warfarin); Optum Clinformatic- Apixaban vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.39 to 0.66]
Statistical Analysis 8: Comparison: MarketScan - Apixaban vs. Warfarin (Apixaban) vs MarketScan - Apixaban vs. Warfarin (Warfarin); MarketScan-Apixaban vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.49 to 0.68]
Statistical Analysis 9: Comparison: Optum Clinformatics - Apixaban vs. Warfarin (Apixaban) vs Optum Clinformatics - Apixaban vs. Warfarin (Warfarin) vs MarketScan - Apixaban vs. Warfarin (Apixaban) vs MarketScan - Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.49 to 0.64]

3. Secondary Outcome: Stroke or Systemic Embolism
Description: The rate of stroke (hemorrhagic, ischemic or stroke of uncertain classification ) or systemic embolism in patients matched on propensity scores and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. For outcome definitions please refer the descriptions section of outcome 4 (Systemic embolism), outcome 5 (Ischemic stroke), outcome 6 (Hemorrhagic stroke) and outcome 7 (Stroke uncertain classification).
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Groups:
- Dabigatran vs. Warfarin (Dabigatran): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of dabigatran, during October 2010 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database or MarketScan before treatment initiation and matched on propensity scores with warfarin
- Dabigatran vs. Warfarin (Warfarin): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of warfarin, during October 2010 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database or MarketScan before treatment initiation and matched on propensity scores with dabigatran
- Rivaroxaban vs. Warfarin (Rivaroxaban): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of rivaroxaban, during July 2011 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database or MarketScan before treatment initiation and matched on propensity scores with warfarin
- Rivaroxaban vs. Warfarin (Warfarin): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of warfarin, during July 2011 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database or MarketScan before treatment initiation and matched on propensity scores with rivaroxaban
- Apixaban vs. Warfarin (Apixaban): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of apixaban, during January 2013 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database or MarketScan before treatment initiation and matched on propensity scores with warfarin
- Apixaban vs. Warfarin (Warfarin): Patients with non- valvular atrial fibrillation (NVAF) and new initiators of warfarin, during January 2013 to September 2015 who were enrolled for a minimum of 12 months in Optum Clinformatics database or MarketScan before treatment initiation and matched on propensity scores with apixaban
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 0.92 [0.77 to 1.08] | 1.13 [0.95 to 1.33] | 1.00 [0.85 to 1.15] | 1.29 [1.11 to 1.50] | 0.81 [0.63 to 1.02] | 1.36 [1.10 to 1.66]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.69 to 1.11]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.66 to 1.02]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.47 to 0.88]

4. Secondary Outcome: Systemic Embolism
Description: The rate of systemic embolism in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. The outcome definition includes following: ICD-9 Diagnoses: 444.x Arterial embolism.
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 0.23 [0.17 to 0.32] | 0.14 [0.08 to 0.22] | 0.21 [0.15 to 0.29] | 0.22 [0.15 to 0.32] | 0.05 [0.02 to 0.11] | 0.17 [0.09 to 0.29]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 1.85, 95% CI 2-sided [1.03 to 3.30]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.65 to 1.71]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.31, 95% CI 2-sided [0.10 to 0.96]

5. Secondary Outcome: Ischemic Stroke
Description: The rate of ischemic stroke in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. The outcome definition includes following: As primary ICD-9 discharge diagnosis (Dx): 433.x1 Occlusion and stenosis of precerebral arteries with cerebral infarction, ICD-9 Dx 434.x1 Occlusion and stenosis of cerebral arteries with cerebral infarction
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 0.63 [0.51 to 0.76] | 0.80 [0.65 to 0.97] | 0.63 [0.52 to 0.75] | 0.90 [0.75 to 1.07] | 0.61 [0.46 to 0.79] | 1.03 [0.80 to 1.29]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.63 to 1.12]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.57 to 0.96]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.45 to 0.94]

6. Secondary Outcome: Hemorrhagic Stroke
Description: The rate of hemorrhagic in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. The outcome definition includes following: As primary ICD-9 discharge diagnosis (Dx): 431.x Intracerebral hemorrhage (ICH)
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 0.07 [0.03 to 0.12] | 0.19 [0.12 to 0.28] | 0.18 [0.12 to 0.25] | 0.18 [0.12 to 0.26] | 0.15 [0.09 to 0.25] | 0.18 [0.10 to 0.31]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.37, 95% CI 2-sided [0.18 to 0.78]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.58 to 1.72]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.38 to 1.87]

7. Secondary Outcome: Stroke Uncertain Classification
Description: The rate of stroke uncertain classification in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. The outcome definition includes following: As primary ICD-9 discharge diagnosis (Dx): ICD-9 Dx code 436.x (acute, but ill-defined cerebrovascular disease).
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.01] | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.04]

8. Secondary Outcome: Major Intracranial Bleeding
Description: The rate of major intracranial bleeding in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. The outcome definition includes following: ICD-9 diagnosis: 430.x Subarachnoid hemorrhage (SAH), 431.x Intracerebral hemorrhage (ICH), 432.x other and unspecified intracranial hemorrhage including 432.1x - subdural hemorrhage
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 0.21 [0.15 to 0.30] | 0.58 [0.46 to 0.73] | 0.44 [0.35 to 0.55] | 0.66 [0.53 to 0.81] | 0.45 [0.32 to 0.60] | 0.69 [0.51 to 0.92]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.39, 95% CI 2-sided [0.25 to 0.59]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.51 to 0.95]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.67, 95% CI 2-sided [0.43 to 1.03]

9. Secondary Outcome: Major Extra-cranial Bleeding
Description: The rate of major extracranial bleeding (Major upper GI bleed, major lower and unspecified GI bleed, major urogenital bleed, major other bleed) in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. For outcome definitions please refer the descriptions section of outcome 11 (Major upper gastrointestinal bleeding), outcome 12 (Major lower gastrointestinal bleeding), outcome 13 (Major urogenital bleeding) and outcome 14 (Other major bleeding).
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 3.78 [3.48 to 4.10] | 5.37 [4.96 to 5.79] | 6.31 [5.94 to 6.69] | 6.54 [6.11 to 6.99] | 3.51 [3.13 to 3.92] | 6.92 [6.31 to 7.58]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.67 to 0.84]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.97 to 1.16]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.47 to 0.63]

10. Secondary Outcome: Major Gastrointestinal (GI) Bleeding
Description: The rate of major gastrointestinal (GI) bleeding (Major upper GI bleeding, major lower/unspecified GI bleeding) in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. For outcome definitions please refer the descriptions section of outcome 11 (Major upper gastrointestinal bleeding) and outcome 12 (Major lower gastrointestinal bleeding).
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 2.39 [2.15 to 2.65] | 2.82 [2.53 to 3.13] | 3.82 [3.53 to 4.12] | 3.43 [3.13 to 3.76] | 1.99 [1.70 to 2.30] | 3.59 [3.16 to 4.07]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.77 to 1.04]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 1.21, 95% CI 2-sided [1.07 to 1.36]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.59, 95% CI 2-sided [0.48 to 0.72]

11. Secondary Outcome: Major Upper Gastrointestinal Bleeding
Description: The rate of Major upper gastrointestinal bleeding in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. The outcome definition includes following: ICD-9 diagnoses: 531.0x, 531.2x, 531.4x, 531.6x, 532.0x, 532.2x, 532.4x, 532.6x, 533.0x, 533.2x, 533.4x, 533.6x, 534.0x, 534.2x, 534.4x, 534.6x, 578.0 OR ICD-9 procedure code 44.43 (endoscopic control of gastric or duodenal bleeding) OR Current Procedural Terminology (CPT) code 43255 (upper gastrointestinal endoscopy including esophagus, stomach, and either the duodenum and/or jejunum as appropriate with control of bleeding, any method).
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 0.51 [0.41 to 0.64] | 0.90 [0.74 to 1.08] | 0.99 [0.85 to 1.15] | 0.88 [0.73 to 1.05] | 0.64 [0.49 to 0.83] | 0.89 [0.68 to 1.14]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.44 to 0.80]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [0.98 to 1.57]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.54 to 1.14]

12. Secondary Outcome: Major Lower Gastrointestinal Bleeding
Description: The rate of lower gastrointestinal bleeding in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. The outcome definition includes following: Lower GI/unspecified GI site bleeds :Diverticulosis of small intestine with hemorrhage: 562.02, Diverticulitis of small intestine with hemorrhage: 562.03, Diverticulosis of colon with hemorrhage: 562.12, Diverticulitis of colon with hemorrhage: 562.13, Hemorrhage of rectum and anus: 569.3x, Angiodysplasia of intestine with hemorrhage: 569.85, Blood in stool: 578.1x, Hemorrhage of GI tract, unspecified: 578.9
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 2.18 [1.96 to 2.43] | 2.48 [2.21 to 2.77] | 3.40 [3.13 to 3.69] | 3.09 [2.80 to 3.39] | 1.61 [1.36 to 1.90] | 3.17 [2.76 to 3.62]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.93, 95% CI 2-sided [0.79 to 1.08]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [1.05 to 1.35]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.44 to 0.67]

13. Secondary Outcome: Major Urogenital Bleeding
Description: The rate of major urogenital bleeding in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. The outcome definition includes following: ICD-9 diagnoses: Hematuria: ICD-9 Dx: 599.7, Excessive/frequent menstruation: ICD-9 Dx 626.2x and secondary diagnosis indicating acute bleeding: anemia (280.0, 285.1, 285.9). Across databases, only one event for dabigatran versus no event among warfarin initiators observed. Across database, four events for rivaroxaban versus no event among warfarin initiators observed. Across database, no events for apixaban and warfarin observed. Therefore HR estimate is not possible.
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 0.01 [0.00 to 0.03] | 0.00 [0.00 to 0.02] | 0.02 [0.01 to 0.06] | 0.00 [0.00 to 0.02] | 0.00 [0.00 to 0.03] | 0.00 [0.00 to 0.04]

14. Secondary Outcome: Other Major Bleeding
Description: The rate of Other major bleeding in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. The outcome definition includes following: Other major bleeds: Hemathrosis: 719.1x, Hemopericardium: 423.0x, Hemoptysis: 786.3x, Epistaxis: 784.7x, Hemorrhage not specified 459.0x, Acute posthemorrhagic anemia 285.1x
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 2.32 [2.08 to 2.57] | 3.65 [3.33 to 4.01] | 4.33 [4.02 to 4.65] | 4.59 [4.24 to 4.97] | 2.54 [2.22 to 2.90] | 4.86 [4.35 to 5.41]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.59 to 078]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.93 to 1.16]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.56, 95% CI 2-sided [0.47 to 0.67]

15. Secondary Outcome: Transient Ischemic Attack (TIA)
Description: The rate of Transient Ischemic Attack (TIA) in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. The outcome definition includes following: ICD-9 Dx code 435.xx (transient cerebral ischemia) as the principal (primary) discharge diagnosis
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 0.21 [0.15 to 0.30] | 0.43 [0.32 to 0.56] | 0.26 [0.19 to 0.34] | 0.31 [0.23 to 0.42] | 0.22 [0.14 to 0.34] | 0.32 [0.20 to 0.48]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.34 to 0.82]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.55 to 1.29]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.41 to 1.42]

16. Secondary Outcome: Myocardial Infarction (MI)
Description: The rate of Myocardial infarction (MI) in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. The outcome definition includes following: ICD-9 Dx 410.X (acute myocardial infarction) excluding 410.x2 (subsequent episode of care), as the principal (primary) or the next (secondary) diagnosis AND a length of stay (LOS) between 3-180 days, or death if LOS is < 3 days
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 0.48 [0.38 to 0.60] | 0.60 [0.48 to 0.75] | 0.53 [0.43 to 0.64] | 0.65 [0.52 to 0.80] | 0.57 [0.43 to 0.75] | 0.74 [0.55 to 0.97]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.60 to 1.15]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.63 to 1.14]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.53 to 1.18]

17. Secondary Outcome: Venous Thromboembolism (VTE)
Description: The rate of Venous Thromboembolism (VTE) in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. For outcome definitions please refer the descriptions section of outcome 18 (Deep vein thrombosis (DVT)) and outcome 19 (Pulmonary Embolism (PE)).
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 0.67 [0.55 to 0.81] | 1.14 [0.96 to 1.34] | 1.20 [1.04 to 1.37] | 1.65 [1.45 to 1.88] | 0.57 [0.43 to 0.75] | 1.21 [0.96 to 1.50]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.50 to 0.84]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); This is a pooled analysis involving data from both MarketScan and Optum databases. MarketScan and Optum Clinformatic-Rivaroxaban vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.69 to 1.01]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.53, 95% CI 2-sided [0.37 to 0.76]

18. Secondary Outcome: Deep Vein Thrombosis (DVT)
Description: The rate of DVT in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. The outcome definition includes following: Validated algorithm: ICD-9 451.1x, ICD-9 451.2x,ICD-9 451.81, ICD-9 451.9x, ICD-9 453.1x, ICD-9 453.2x, ICD-9 453.8x, ICD-9 453.9x ; Not in the validated algorithm but will be included following Mini-Sentinel recommendation for VTE outcome: ICD-9 453.40 (Venous embolism and thrombosis of unspecified deep vessels of lower extremity (includes DVT), ICD-9 453.41 (Venous embolism and thrombosis of deep vessels of proximal lower extremity (includes femoral, iliac, popliteal, thigh, and upper leg), ICD-9 453.42 (Venous embolism and thrombosis of deep vessels of distal lower extremity (includes calf, lower leg, peroneal, and tibia), ICD-9 453.0 (Hepatic vein thrombosis)
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 0.46 [0.36 to 0.58] | 0.78 [0.64 to 0.95] | 0.78 [0.66 to 0.93] | 1.09 [0.93 to 1.28] | 0.41 [0.29 to 0.56] | 0.75 [0.57 to 0.99]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 3]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.65, 95% CI 2-sided [0.47 to 0.88]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.65 to 1.04]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.39 to 0.92]

19. Secondary Outcome: Pulmonary Embolism (PE)
Description: The rate of Pulmonary Embolism (PE) in patients who are matched on propensity score and calendar quarter of initiation. Event rates were calculated as the total number of patients in each treatment group who had the outcome during follow-up divided by the total person-years at risk in the cohort. The outcome definition includes following: ICD-9 415.1x (pulmonary embolism and infarction)
Time Frame: From October 2010 to September 2015 (the study period)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Incidence rate per 100 person-years
Arm/Group | Dabigatran vs. Warfarin (Dabigatran) | Dabigatran vs. Warfarin (Warfarin) | Rivaroxaban vs. Warfarin (Rivaroxaban) | Rivaroxaban vs. Warfarin (Warfarin) | Apixaban vs. Warfarin (Apixaban) | Apixaban vs. Warfarin (Warfarin)
Number analyzed (Participants) | 29448 | 29448 | 35520 | 35520 | 19588 | 19588
Incidence rate per 100 person-years | 0.29 [0.21 to 0.38] | 0.46 [0.35 to 0.59] | 0.54 [0.44 to 0.66] | 0.81 [0.67 to 0.97] | 0.22 [0.14 to 0.34] | 0.62 [0.45 to 0.83]
Statistical Analysis 1: Comparison: Dabigatran vs. Warfarin (Dabigatran) vs Dabigatran vs. Warfarin (Warfarin); This is a pooled analysis involving data from both MarketScan and Optum databases. MarketScan and Optum Clinformatic- Dabigatran vs. Warfarin (as reference group); Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.47 to 1.04]
Statistical Analysis 2: Comparison: Rivaroxaban vs. Warfarin (Rivaroxaban) vs Rivaroxaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 6]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.60 to 1.05]
Statistical Analysis 3: Comparison: Apixaban vs. Warfarin (Apixaban) vs Apixaban vs. Warfarin (Warfarin); [analysis description as in outcome 1, analysis 9]; Test type: Other; Regression, Cox; [statistical method as in outcome 1, analysis 3]; Hazard Ratio (HR) = 0.42, 95% CI 2-sided [0.24 to 0.73]

ADVERSE EVENTS:
Time Frame: Individual safety reporting was not applicable for this study
Description: This was an observational study based on existing data (secondary data use); all patient data are de-identified and analyzed in aggregate. Individual patient safety related information was not captured during this study; therefore the individual safety reporting was not applicable for this study.
Arm/Group | Optum Clinformatics - Dabigatran | Optum Clinformatics - Warfarin | Optum Clinformatics - Rivaroxaban | Optum Clinformatics - Apixaban | MarketScan - Dabigatran | MarketScan - Warfarin | MarketScan - Rivaroxaban | MarketScan - Apixaban
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT02081807/Prot_SAP_000.pdf